CLINICAL TRIAL: NCT00010842
Title: Natural Antioxidants in the Treatment of Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000066-01P1 (NIH); P50AT000066-01 (NIH); NCT00009438 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ginkgo Extract; Thioctic Acid; Fatty Acids, Essential

INTERVENTIONS:
Drug: Ginkgo biloba
Drug: Alpha-lipoic acid
Drug: Vitamin E/Selenium
Drug: Essential fatty acids

SUMMARY:
The purpose of this study is to compare the effectiveness of three antioxidant regimens in treating the symptoms of multiple sclerosis (MS).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an immune mediated disease of the central nervous system that affects over 350,000 Americans. T lymphocytes, macrophages and soluble mediators of inflammation cause demyelination and axonal injury in MS. Activated macrophages release nitric oxide and oxygen free radicals that cause demyelination and axonal injury in MS and experimental autoimmune encephalomyelitis (EAE). Natural antioxidants may favorably influence the course of MS by decreasing oxidative injury. Chronic relapsing EAE in mouse models is clinically and pathologically useful for testing potential therapies for MS.

This study will assess three natural antioxidant regimens for their potential as treatments for MS: Ginkgo biloba, alpha-lipoic acid/essential fatty acids, and vitamin E/selenium. The effects of each regimen will be compared to determine which regimen appears most effective at suppressing EAE and decreasing markers of oxidative injury in patients with MS. As part of this study, two smaller trials will be conducted. A Phase I/II trial in patients with MS will determine if the selected antioxidant regimen can decrease disease activity as detected with gadolinium-enhanced magnetic resonance imaging. The results of this study will serve as the basis for a Phase III trial to assess the long term effectiveness of natural antioxidant therapy in MS.

ELIGIBILITY:
Exclusion Criteria:

* Pregnant
* Other significant health problems

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dennis Bourdette, Principal Investigator — VA Medical Center-Brooklyn
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States